CLINICAL TRIAL: NCT02500784
Title: Improving Beta-2 Adrenergic Signaling in Alzheimer's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ran out before study started, prior PI left institution.
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Alzheimer's Association (Other); Mylan Inc. (Industry)
Responsible Party: Principal Investigator, J. Wesson Ashford, Clinical Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASJ0015
Record Dates: First submitted 2015-05-19; First posted 2015-07-17 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease; Cognitive Dysfunction
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Formoterol A (Active Comparator): 12 months, formoterol, 20microgram/2ml, inhaler, BID
  Interventions: Drug: Formoterol A
- Formoterol B (Placebo Comparator): 12 months, normal saline, 2ml, inhaler, BID
  Interventions: Other: Formoterol B (placebo)

INTERVENTIONS:
Drug: Formoterol A — 20mg/2mL, BID inhaler for 12 months: until progression or unacceptable toxicity develops.
  Other Names: Performist
  Arms: Formoterol A
Other: Formoterol B (placebo) — 2mL, BID inhaler for 12 months
  Arms: Formoterol B

SUMMARY:
The purpose of this study is to test the effects of long-term therapeutic doses of formoterol, on a) cerebrospinal fluid (CSF) tau levels, and Amyloid Beta protein 40/42 levels in the CSF, and b) cognitive function in people with mild to moderate Alzheimer' Disease (AD).

DETAILED DESCRIPTION:
The purpose of this study is to test the effects of long-term therapeutic doses of formoterol, on a) cerebrospinal fluid CSF tau levels, and A-beta amyloid protein 40/42 levels, and b) cognitive function: NE-ergic neurons undergo significant degeneration in AD. This system plays a significant role in cognition. Recent studies have indicated that increasing NE levels in the brain would significantly improve microglia migration and clearance of A-beta amyloid protein 40/42 levels in mouse models of AD. The investigators plan to test whether long- term daily treatment with inhaled formoterol solution would improve the structure and function of hippocampal neurons in AD. Study Design: Randomization and initiation of experimental treatment: All participants will be given formoterol daily for 52 weeks. The active regimen will be initiated as (20 micro gram, BID). The dose will be decreased if there is evidence of side effects, including cardiac or respiratory alteration changes, gastro-intestinal disturbances or neurological issues.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 50-85,
* Mild-to-moderate AD (NINCDS/ADRDA criteria for probable AD will be used to establish AD diagnosis).
* MMSE 16-26.

Exclusion Criteria:

* Non-AD dementia or significant neurological disease such as Parkinson's disease, stroke, brain tumor,multiple sclerosis, seizure disorder, focal brain lesion, or head injury with loss of consciousness.
* Hypothyroidism, congestive heart failure (New York Heart Association Class III or IV), significant extrapyramidal symptoms on neurological examination, serum creatinine>1.3 mg/dl, significant arrhythmias or conduction defect abnormalities on ECG,
* Use of another beta2 adrenergic drug within the last 2 months.
* Residence in a long-term care facility.
* Evidence of any significant clinical disorder or laboratory finding that renders the person unsuitable for receiving an investigational new drug.
* Known hypersensitivity or prior exposure to formoterol.
* Active asthma or family history of asthma.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cognition Evaluation | 1 Month
  Participants will be administered the CANTAB every month for 16 months
Brain-derived neurotrophic factor (BDNF) Evaluation | Baseline and month 16
  Samples of Plasma and Cerebral Spinal Fluid Biomarkers will be taken at baseline and month 16

SECONDARY OUTCOMES:
Amyloid accumulation | Baseline and month 16
  Molecular Imaging will be taken at baseline and month 16

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Salehi, M.D.,Ph.D., Principal Investigator — Stanford Medical School
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No subjects enrolled